CLINICAL TRIAL: NCT00336115
Title: Safety and Immunogenicity of Adult Formulation Tetanus and Diphtheria Toxoids Adsorbed Combined With Acellular Pertussis (Tdap) Vaccine Following Blood and Morrow Transplantation in Adults
Brief Title: The Safety and Immunogenicity of Acellular Pertussis Vaccine in Bone Marrow Transplant Recipients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Queen Elizabeth II Health Sciences Centre (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: qeii
Record Dates: First submitted 2006-06-09; First posted 2006-06-12 (Estimated); Last update posted 2007-10-23 (Estimated); Status verified 2007-10

CONDITIONS: Pertussis
Keywords: pertussis; bone marrow transplant
MeSH Terms: conditions — Whooping Cough | interventions — Tetanus Toxoid; adacel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Tetanus and Diphtheria Toxoids Adsorbed Combined with Acellular Pertussis (Adacel)

SUMMARY:
The purpose of this study is to determine if pertussis (whooping cough) vaccine is safe and produces an appropriate immune response against pertussis in blood and marrow transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-64
* BMT at the QEII Health Sciences Centre
* BMT within last 12 months
* Able to read and write English language
* Able to give consent

Exclusion Criteria:

* Active infection
* Active GVHD
* Recent IVIG
* Allergy to components of vaccine
* Diphtheria or tetanus vaccination within 18 months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-07; Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
Safety of the vaccine | 28 days post-dose

SECONDARY OUTCOMES:
Immunogenicity of vaccine | 60 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Monique L MacFarlane Conrad, MSc, Principal Investigator — Dalhousie University Medical School; Shelly McNeil, MD, Study Director — Queen Elizabeth II Health Sciences Centre